CLINICAL TRIAL: NCT03399305
Title: Safety and Efficacy of Apixaban in Severe Renal Impairment
Status: Withdrawn | Type: Observational
Why Stopped: investigators have decided not to continue with the study
Sponsor: Albert Einstein College of Medicine (Other)
Responsible Party: Principal Investigator, Henny Billett, Chief of Hematology, Albert Einstein College of Medicine
Other Study IDs: 2017-7774
Record Dates: First submitted 2018-01-08; First posted 2018-01-16 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Renal Disease, End Stage; Anticoagulant-induced Bleeding
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Despite emergence of new anticoagulants over the last few years, patients with advanced chronic kidney disease still have limited options and are usually managed with warfarin after venous thromboembolism or diagnosis of atrial fibrillation. The use of all direct oral anticoagulants is not recommended in patients with creatinine clearance below 15 mL/min. Apixaban has the lowest fraction of renal excretion (27%) and is sometimes used in patients with CKD V (GFR < 15 mL/min/BSA) and end stage renal disease (ESRD). Until recently, data on apixaban use in this population were limited to pharmacodynamics as patients with severe renal impairment were excluded from clinical trials. In a 2016 study, it was found that ESRD resulted in 36% increase in apixaban AUC but no increase in Cmax, and that hemodialysis had a limited impact on apixaban clearance.1 There are now data available on inpatient use of apixaban vs.coumadin in patients with creatinine clearance below 25 ml/min.2 There was no significant difference in bleeding events between the two groups but the study period was limited to a hospital admission and may not reflect bleeding risk of long-term anticoagulation.

Use of warfarin in patients on hemodialysis entails several disadvantages in this population. The need for INR monitoring adds clinic visits for patients that already spend a great portion of their time in healthcare facilities. Numerous drug interactions, involving warfarin, complicate management of ESRD patients that are often on many medications. The reduced risk of intracranial bleeding on apixaban, compared to warfarin, in the ARISTOTLE study, is an important consideration in patients that may already be at increased risk due other factors such as uremia and concurrent antiplatelet agents.

DETAILED DESCRIPTION:
This is a retrospective cohort study. The investigators will use Clinical Looking Glass (CLG) to identify all adult patients with creatinine clearance < 15 ml/min who were treated with apixaban or warfarin, for at least 1 month, between 3/1/2013 and 3/1/2017. The investigators will then review electronic charts in Carecast and Epic to gather data about bleeding and thrombotic events.Primary outcome: clinically significant bleeding, per Control of Anticoagulation Subcommittee criteria: 1) fatal bleed; 2) symptomatic bleed at anatomically critical sites such as intracranial, intraspinal, intraocular, or pericardial hemorrhage; 3)symptomatic noncritical bleeds resulting in transfusion of 2 units or more of red blood cells or drop in hemoglobin of at least 2.0 g/dl.4 Secondary outcomes: venous thromboembolism, cerebrovascular accident, intracranial hemorrhage, bleeding related to HD access

ELIGIBILITY:
Inclusion Criteria:

* Patients with creatinine clearance <15 mL/min who are on anticoagulation with apixaban or warfarin.

Exclusion Criteria:

* Patients without end stage renal disease who are not on anticoagulation with apixaban or warfarin.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with creatinine clearance <15 mL/min who are on anticoagulation with apixaban or warfarin.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-05-10 (Actual); Primary Completion 2019-07-07 (Actual); Study Completion 2022-08-24 (Actual)

PRIMARY OUTCOMES:
Clinically significant bleeding | 4 years
  1) fatal bleed; 2) symptomatic bleed at anatomically critical sites such as intracranial, intraspinal, intraocular, or pericardial hemorrhage; 3) symptomatic noncritical bleeds resulting in transfusion of 2 units or more of red blood cells or drop in hemoglobin of at least 2.0 g/dl

CONTACTS AND LOCATIONS:
Overall Officials: Henny H Billett, MD, Principal Investigator — Albert Einstein College of Medicine and Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No